CLINICAL TRIAL: NCT02680340
Title: Longterm Clinical Outcome Study of the Femoral Cementless Ti/HA Polarstem - A Multicenter Retrospective 10-years Follow-up Study
Brief Title: POLARSTEM Retrospective Multicenter Study
Acronym: PR
Status: Completed | Type: Observational
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Other Study IDs: 14-4562-05
Record Dates: First submitted 2016-01-05; First posted 2016-02-11 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Osteoarthritis
Keywords: Total Hip Arthroplasty THA
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Total Hip Arthroplasty — Patients who had a primary THA between 2002 and 2005
  Other Names: Polarstem primary THA

SUMMARY:
The primary purpose of this study is to demonstrate the POLARSTEM™ Ti/HA cumulative femoral stem revision rate at 10 years.

The secondary purpose of this study is to provide 10 years of safety and effectiveness data of POLARSTEM™ Ti/HA in terms of radiographic and clinical performance

DETAILED DESCRIPTION:
This is a multicenter retrospective longterm clinical outcome study conducted in up to 6 hospitals in France. 502 subjects who have undergone THA with POLARSTEM™ from 2002 to 2005 will be enrolled in this study and clinical and radiographically followed up for at least 10 years. Subjects who have not reached the 10-year post surgery timepoint will be invited to a 10-year post-operative follow-up visit to obtain the clinical and radiographic outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Subject required and received primary total hip arthroplasty between 2002 and 2005.
2. Subject received the POLARSTEM™ Ti/HA unilateral or bilateral, due to severe hip joint damage resulting from arthrosis, degenerative disease, traumatic events, inflammatory or rheumatoid processes.
3. Subject received the non-cemented POLARSYSTEM (POLARSTEM™ Ti/HA in combination with POLARCUP™).
4. Subject was aged between 18 and 75 at time of surgery.
5. Signed Informed Consent (ICF).

Exclusion Criteria:

1. Subject received the cemented POLARSTEM™.
2. Previously failed endoprosthesis and/or THR components in relevant hip.
3. Medical or mental health conditions which could impair the stubject's ability or willingness to comply with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 502 male and female subjects who have undergone THA with POLARSTEM™ from 2002 to 2005 will be enrolled in this study and clinical and radiographically followed up for at least 10 years.
Sampling Method: Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Femoral stem revision rate at 10 years for any reason | since surgery until 10 years Follow Up
  Long term cumulative femoral stem revision rate of Polarstem will be evaluated in 502 subjects

SECONDARY OUTCOMES:
Number of subjects with revision of any components for any reason | date of surgery until 10 years Follow Up
  Long-term cumulative revision rate of the cup will be evaluated in 502 subjects
Standard radiographic assessment at least at 10 years | date of surgery and at 10 years Follow Up
  radiographic evaluation on x-rays to assess the osseointegration and orientation of cup and stem, heterotopic ossification, signs of radiolucent lines, osteolysis, atrophy and hypertrophy
Hip Disability and Osteoarthritis Outcome Score (HOOS) at least at 10-year assessment as patient reported outcome (PRO | at 10 years Follow Up
Merle D'Aubigné and Postel (MAP) at least at 10-year assessment | pre-operative and at 10 years Follow Up
Adverse Events | through study completion, an average of 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Fiquet, Dr. med., Principal Investigator — Infirmerie Protestante de Lyon
Locations (5):
- France (5):
  - Clinique la Parisière, Bourg-de-Péage
  - Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - Centre Hospitalier du Forez- Montbrison, Montbrison
  - Centre Hospitalier de Montélimar, Montélimar
  - Clinique du Renaison, Roanne

IPD SHARING:
Plan to Share IPD: No